CLINICAL TRIAL: NCT05871060
Title: Effect of a Novel Protein Supplement on Appetite in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Principal Investigator, Katy Horner, Lecturer in Sport and Exercise Science, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LS-22-64-Horner; TC201800025 (Other Grant/Funding Number: Food for Health Ireland)
Record Dates: First submitted 2023-03-31; First posted 2023-05-23 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Aging; Appetite Loss
Keywords: Appetite; Poor Appetite; Ageing; Whey protein hydrolysate; Visual analogue scale; Energy intake; Ghrelin
MeSH Terms: conditions — Anorexia | interventions — Whey

STUDY DESIGN:
Intervention Model Description: All participants undertake all three experimental conditions in a random order.
Who Masked: Participant, Investigator
Masking Description: Out of three treatments, the investigator is blinded for two of them (pre-labelled as A and B).
  The participant is fully blinded, i.e. treatments will be served in black cups and vanilla-flavoured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- whey concentrate supplement (Active Comparator): 2,2 grams of whey concentrate dissolved in 100 mL of water
  Interventions: Dietary Supplement: Whey Protein Concentrate
- whey hydrolysate supplement (Experimental): 2,2 grams of whey hydrolysate dissolved in 100 mL of water
  Interventions: Dietary Supplement: Whey hydrolysate
- still flavoured water (Placebo Comparator): 100 mL of vanilla-flavoured water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey Protein Concentrate — Whey protein concentrate consumed 30 minutes prior to breakfast and lunch meals
  Arms: whey concentrate supplement
Dietary Supplement: Placebo — Flavoured water consumed 30 minutes prior to breakfast and lunch meals
  Arms: still flavoured water
Dietary Supplement: Whey hydrolysate — Whey hydrolysate consumed 30 minutes prior to breakfast and lunch meals
  Arms: whey hydrolysate supplement

SUMMARY:
An acute randomized crossover trial comparing the effects of the whey hydrolysate, whey protein concentrate and placebo (still flavored water) on appetite and energy intake in older adults. Both low-dose whey-derived treatment and placebo will be administered 30 minutes prior to breakfast and lunch meals. Moreover, ghrelin secretion and activity will be monitored throughout the morning until the lunch time. Appetite will be assessed through visual analogue scale questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling,
* Age 60+ years
* Poor appetite (Simplified Nutritional Appetite Questionnaire (SNAQ) score </=14, answer a, b or c to Q.1 on SNAQ or answer b, c, or d to CES-D question regarding poor appetite in the past week)
* BMI 20-25kg/m2

Exclusion Criteria:

1. Current medical condition or medication known to impact appetite or energy intake
2. Other medical condition that would impact study participation and outcomes, as judged by the study investigator.
3. Heavy smoker (>10/day)
4. Inability to come to study centre
5. Currently participating in another intervention study
6. Lacking informed consent
7. Allergic to or unwilling to consume any of the study test foods
8. Loss of taste or smell associated with COVID-19
9. Unable to walk across a room

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Pre-meal and changes in Composite Appetite Score | 8.5 hours: fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes after ingestion of supplement and a standard meal; at 30, 60, 120 and 180 minutes following ingestion of supplement and lunch test meal. And immediately after each test meal.
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess appetite, at fourteen (14) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score is derived from VAS ratings of hunger, fullness, desire to eat and prospective food consumption.
Energy intake (EI) (kilocalories) | 24 hours from breakfast, lunch and dinner meals, as well as from evening and night from provided snackbox.
  24-hour energy intake measurement. Participants will be served a standardised fixed breakfast and ad libitum lunch and dinner meals in the laboratory and provided with an evening snack box. 24 hour EI (kilocalories) will be measured objectively, by weighing foods before and after consumption and calculating energy intake based on their nutritional data. Total accumulated energy intake includes standard breakfast meal, ad libitum lunch meal, ad libitum dinner meal and bag with known foods for the evening time.

SECONDARY OUTCOMES:
Palatability - Pleasantness | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Filling | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Satisfaction | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Taste | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Sweet | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Savoury | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  100 millimetre Visual Analogue Scales (VAS) will be used after each test meal: breakfast, lunch and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Pre-meal and changes in glucose | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in insulin | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in growth hormone | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in cortisol | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in GLP-1 | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in PYY | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Total Ghrelin | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Acylated Ghrelin | 4 hours, from fasting state (morning) to immediately prior to lunch meal (afternoon): fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Hunger | 8.5 hours: fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement and a standard meal; at 30, 60, 120 and 180 minutes following ingestion of supplement and test meal.
  Validated 100 mm Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at fourteen (14) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the extreme positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score derived from aspects such as hunger, fullness, desire to eat and prospective food consumption will be calculated. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Fullness | 8.5 hours: fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement and a standard meal; at 30, 60, 120 and 180 minutes following ingestion of supplement and test meal.
  Validated 100 mm Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at fourteen (14) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the extreme positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score derived from aspects such as hunger, fullness, desire to eat and prospective food consumption will be calculated. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Desire to Eat | 8.5 hours: fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement and a standard meal; at 30, 60, 120 and 180 minutes following ingestion of supplement and test meal.
  Validated 100 mm Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at fourteen (14) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the extreme positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score derived from aspects such as hunger, fullness, desire to eat and prospective food consumption will be calculated. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Prospective Food Consumption | 8.5 hours: fasting, before breakfast, at 30, 60, 120, 180 and 210 minutes following ingestion of supplement and a standard meal; at 30, 60, 120 and 180 minutes following ingestion of supplement and test meal.
  Validated 100 mm Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at fourteen (14) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the extreme positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score derived from aspects such as hunger, fullness, desire to eat and prospective food consumption will be calculated. Fasting, mean and AUC values will be calculated.
Liking of test meals | Mean of ratings taken immediately following the three test meals (single measure) - breakfast, lunch and dinner
  9-point likert scale from 0 dislike extremely to 9 like extremely

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland